CLINICAL TRIAL: NCT05452720
Title: MASA Valve Early Feasibility Study
Acronym: MVEFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PECA Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: G220040
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Tetrology of Fallot; Pulmonary Stenosis; Truncus Arteriosus; Transposition of Great Vessels; Pulmonary Atresia; Ross Procedure
Keywords: Right Ventricular Outflow Tract Reconstruction; Pulmonary Valve; MASA Valve; Pulmonary Valve Replacement
MeSH Terms: conditions — Tetralogy of Fallot; Pulmonary Valve Stenosis; Truncus Arteriosus, Persistent; Transposition of Great Vessels; Pulmonary Atresia

STUDY DESIGN:
Intervention Model Description: The MASA Valve Early Feasibility Study (MVEFS) is a multi-center, non-randomized, prospective, interventional clinical study to determine the safety and probable benefit of MASA Valve pulmonary valved conduit in the indicated subset of patients requiring Right Ventricular Outflow Tract Reconstruction (RVOTR).
  Each implanted subject will be consented to be followed for a total of 5 years with a post-op, 30 day (30+7), 180 day (180±30) and 1 year follow-up (365 ± 90 days) followed by an annual follow up until 5 years (annual visits with a window of ± 90 days per visit), or until trial closure. Total expected duration of the trial is approximately 5 year from the last enrolled patient. Intermediary results of the trial may be calculated prior to completion of the 1-year (365 ± 90 days) endpoint of all patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental Arm (Experimental): This is a single-arm study. All participants in this study will undergo implantation with MASA Valve.
  Interventions: Device: Surgical Right Ventricular Outflow Tract Reconstruction

INTERVENTIONS:
Device: Surgical Right Ventricular Outflow Tract Reconstruction — Surgical replacement of the Pulmonary Valve or a previously implanted prosthetic with the investigational device (MASA Valve)

SUMMARY:
The MASA Valve Early Feasibility Study (MVEFS) multi-site interventional clinical trial within the United States of America with each center following a common protocol.The objective of the trial is to evaluate the safety and probable benefit of MASA Valve in the indicated subset of patients requiring Right Ventricular Outflow Tract Reconstruction (RVOTR). As an early feasibility study, the purpose is determine the feasibility of success of the device in order to gather early data towards a future pivotal study and/or regulatory clearance submission.

DETAILED DESCRIPTION:
The MASA Valve is a bi-leaflet pulmonary valved conduit. The MASA Valve has an ePTFE conduit and ePTFE leaflets fixtured to the conduit with polypropylene suture. The device has a pad-printed design on the outer conduit surface indicating the valve position and direction of flow. .

The MASA Valve is intended to be used to reconstruction the Right Ventricular Outflow Tract (RVOT) and provide a functional pulmonary valve. Once implanted, the MASA Valve provides a pathway for blood from the Right Ventricle (RV) to the Pulmonary Arteries (PAs), while the integrated valve helps to prevent backflow into the RV. The MASA Valve Indications for Use are:

The MASA Valve pulmonary valved conduit is indicated for correction or reconstruction of the right ventricular outflow tract (RVOT) in patients aged less than 22 years with any of the following congenital cardiac malformations:

* Pulmonary Stenosis
* Tetralogy of Fallot
* Truncus Arteriosus
* Transposition of Great Vessels
* Pulmonary Atresia

In addition, the MASA Valve is indicated for the replacement of previously implanted, but dysfunctional, pulmonary valves, valved conduits or conduits, as well as for use in the Ross Procedure when the native RVOT is being used to reconstruct the Aorta.

Treatments currently available for the above-stated conditions include biologic-tissue-based valved conduits (Homografts and Contegra Glutaraldehyde-fixed Bovine Jugular Vein), Intra-operatively constructed valved conduits made from off-the-shelf vascular grafts and cardiovascular membranes, and non-valved cardiovascular conduits. Based on existing evidence it is believed the potential benefits of MASA Valve outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

1. At least one of the following: Right Ventricular to Pulmonary Artery mean gradient > 35mm Hg, moderate or severe Pulmonary regurgitation (≥3+), or clinical indication for replacement of their native or prosthetic pulmonary valve with a prosthesis.
2. Age < 22 years
3. Patient is geographically stable and willing to return for 1 year follow-up for the trial.
4. Patient's legal guardian should be willing to provide informed consent (IC) at the hospital location where they are being enrolled.
5. The patient, and the patient's parent / legal representative where appropriate, and the treating physician agree that the subject will return for all required post-procedure follow up visits and the subject will comply with clinical investigation plan required follow-up visits.

Exclusion Criteria:

1. Patient is in need of or has presence of a prosthetic heart valve at any other position
2. Patient has a need for concomitant surgical procedures (non-cardiac)
3. Patients with previously implanted pacemaker (including defibrillators) or mechanical valves
4. Patient has an active bacterial or viral infection or requiring current antibiotic therapy (if temporary illness, patient may be a candidate 4 weeks after discontinuation of antibiotics)
5. Patient has an active endocarditis
6. Leukopenia, according to local laboratory evaluation of white blood cell count
7. Acute or chronic anemia, according to local laboratory evaluation of hemoglobin Patients can be transfused to meet eligibility criteria
8. Thrombocytopenia, defined as Platelet count < 150,000/mm3 Patients can be transfused to meet eligibility criteria
9. Severe chest wall deformity, which would preclude placement of the PV conduit
10. Known hypersensitivity to anticoagulants and antiplatelet drugs and to the device materials
11. Immunocompromised patient defined as: autoimmune disease, patients receiving immunosuppressant drugs or immune stimulant drugs
12. Patient has chronic inflammatory / autoimmune disease
13. Need for emergency cardiac or vascular surgery or intervention
14. Major or progressive non-cardiac disease (liver failure, renal failure, cancer) that has a life expectancy of less than one year
15. Currently participating, or participated within the last 30 days, in an investigational drug or device study
16. Alcohol or drug abuse as defined by DSM IV-TR criteria for substance abuse - this includes the illicit use of cannabis within the last 12 months
17. Patient has medical, social or psychosocial factors that, in the opinion of the Investigator, could have impact on safety or compliance

Ages: 0 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from device related death | 1 year
  Percentage of patients that have not died related to the device 1 year from implantation
Freedom from Explant | 1 year
  Percentage of patients that have not undergone device explant within 1 year from implantation
Freedom from Device-Related Reoperation | 1 year
  Percentage of patients that have not undergone re-operation related to the device within 1 year from implantation
Freedom from Device-Related Catheter Intervention | 1 year
  Percentage of patients that have not undergone device related catheter based intervention within 1 year from implantation
Freedom from Endocarditis | 1 year
  Percentage of patients that have not had endocarditis within 1 year from implantation
Freedom from Thrombus | 1 year
  Percentage of patients that have not had a serious thrombotic event related to the device within 1 year from implantation
Freedom from Major Hemorrhage | 1 year
  Percentage of patients that have not had a major bleeding episode related to the device within 1 year from implantation

SECONDARY OUTCOMES:
Freedom from Moderate or Greater Pulmonary Regurgitation | 1 year
  Percentage of patients that show less than Moderate Pulmonary Regurgitation within 1 year from implantation on Echocardiographic assessment
Freedom from Pulmonary Gradient ≥36mmHg | 1 year
  Percentage of patients that have a Pulmonary Gradient <= 36mmHg within 1 year from implantation on Echocardiographic assessment
Freedom from device valve failure | 1 year
  Percentage of patients that show do not show valve functional failure on Echocardiographic assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Morales, MD, Principal Investigator — Cinncinnati Childrens Hospital
Locations (5):
- United States (5):
  - OSF Childrens Hospital of Illinois, Peoria, Illinois
  - Boston Childrens Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Only anonymized data is intended to be shared with other clinicians.